CLINICAL TRIAL: NCT04920552
Title: Abdominal Binders to Treat Orthostatic Hypotension in Parkinsonian Syndromes: a Randomized, Placebo-controlled, Double-blind, Crossover Phase II Trial
Brief Title: Abdominal Binders to Treat Orthostatic Hypotension in Parkinsonian Syndromes
Acronym: ABOH-PS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinik für Neurologie, Innsbruck (Other)
Responsible Party: Principal Investigator, Gregor Wenning, Head of Division of Neurobiology, Department of Neurology, Medical University of Innsbruck; Principle Investigator; Professor DDr. MD MSc, Universitätsklinik für Neurologie, Innsbruck
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1483/2020
Record Dates: First submitted 2021-05-26; First posted 2021-06-10 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease; Multiple System Atrophy, Parkinson Variant; Orthostatic; Hypotension, Neurogenic
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Hypotension

STUDY DESIGN:
Intervention Model Description: monocentric, randomized, placebo-controlled, double-blind, crossover phase II trial with an open-label treatment extension phase
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo binder first (Placebo Comparator): Participants in this arm will wear the placebo comparator ("Clima Care" body warmer, Bort Medical GmbH) for 2 hours on treatment day-1 (i.e. Visit 1), followed by the active comparator ("ABDO-SYNCRO 3-BAHNIG" elastic abdominal binder, SYNCRO-MED GmbH) for 2 hours on treatment day-2 (i.e. Visit 2).
  Interventions: Device: Elastic abdominal binder; Device: Placebo binder
- Elastic abdominal binder first (Active Comparator): Participants in this arm will wear the active comparator ("ABDO-SYNCRO 3-BAHNIG" elastic abdominal binder, SYNCRO-MED GmbH) for 2 hours on treatment day-1 (i.e. Visit 1), followed by the placebo comparator ("Clima Care" body warmer, Bort Medical GmbH) for 2 hours on treatment day-2 (i.e. Visit 2).
  Interventions: Device: Elastic abdominal binder; Device: Placebo binder

INTERVENTIONS:
Device: Elastic abdominal binder — The "ABDO-SYNCRO 3-BAHNIG" is an elastic abdominal binder with a 3-stripes Velcro fastening, capable of developing a 20 ± 2 mmHg pressure on the abdominal wall. This device will be tested as potentially beneficial with respect to the mentioned primary and secondary outcomes. The investigators anticipate to use this elastic abdominal binder, since participants of a previous trial reported this device to be comfortable enough and to have used it regularly during the open-label follow-up phase. Size will be chosen depending on the abdominal circumference of the participant, according to the size tables provided from the manufacturer (SYNCRO-MED GmbH).
  Other Names: "ABDO-SYNCRO 3-BAHNIG" elastic abdominal binder, SYNCRO-MED GmbH
Device: Placebo binder — "Clima Care" is a simple body warmer, developing maximal 3±2 mmHg pressure on the abdominal wall. This device will be used as placebo comparator of the present clinical trial. Size will be chosen depending on the abdominal circumference of the participant, according to the size tables provided from the manufacturer.
  Other Names: "Clima Care" body warmer, Bort Medical GmbH

SUMMARY:
The purpose of the present clinical trial is to determine whether the use of an elastic abdominal binder is effective in the non-pharmacological management of symptomatic, neurogenic orthostatic hypotension (OH) in individuals suffering from Parkinson's disease (PD) or Parkinson variant multiple system atrophy (MSA-P).

DETAILED DESCRIPTION:
This is a monocentric, randomized, placebo-controlled, double-blind, crossover phase II clinical trial with an open-label treatment extension phase. The investigators plan to recruit n = 30 individuals with MSA-P or PD with known or suspected OH.

At the Screening Visit, after patient information and written informed consent, the participants will first undergo a comprehensive neurological and cardiological evaluation, as well cardiovascular autonomic function testing to confirm the diagnosis of symptomatic, neurogenic OH.

Afterwards, the participants will be asked to wear physical activity monitoring (PAM) sensors for five consecutive days and to measure the blood pressure (BP) regularly following a home BP diary (i.e. Home Phase I).

On treatment day-1 (i.e. Visit 1), the participants will undergo an instrumented in-lab gait analysis, followed by a head-up tilt and active standing test. Afterwards, they will wear the first type of binder for two hours (either the investigational elastic abdominal binder or the placebo-comparator binder, depending on the randomization assignment). At the end of the two hours, the participants will repeat the in-lab gait analysis and the head-up tilt-/active standing test.

After one-day wash-out, the same procedure of treatment day-1 (i.e. Visit 1) will be repeated with the outstanding type of binder (i.e. treatment day-2, Visit 2).

At the end of this, all participants will be invited to wear the investigational elastic abdominal binder and the PAM sensors for five more days and to repeat the home BP measurements (i.e. Home Phase II).

A final follow-up visit is scheduled to return the PAM sensors, the BP monitor and to detect eventual adverse and serious adverse events occurred during Home Phase II.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of possible or probable MSA-P (Gilman 2008) or clinically established PD (Postuma 2015);
* 50 to 85 years of age;
* laboratory-confirmed symptomatic (i.e. OHQ - OH Symptom Assessment item #1 ≥ 4), neurogenic OH at screening visit or previously diagnosed as such (i.e. neurogenic OH ratio [≤ 0.492 Δ heart rate rise/systolic BP fall] or missing BP overshoot at phase IV of Valsalva maneuver;
* stable medication schedule in the preceding 3 weeks;
* no infectious disease in the preceding 3 weeks;
* Hoehn & Yahr stage ≤ 3;
* gait item of the Unified MSA Rating Scale (UMSARS) Part II or the Movement Disorder Society - Unified PD Rating Scale (MDS-UPDRS) Part III score < 3;
* body sway item of the UMSARS II/MDS-UPDRS III score < 3;
* arising from chair item of the UMSARS II/MDS-UPDRS III score < 3;
* full legal capacity;
* written informed consent has been obtained.

Exclusion Criteria:

* participation in other interventional trials;
* prescribed and regular use of abdominal binders OR compression stockings for OH treatment;
* other major neurologic or psychiatric diseases which could influence OH or gait;
* untreated diabetes mellitus with clinical features of peripheral neuropathy;
* non-neurological causes of gait disorders;
* major cardiac diseases (ischemic, structural, arrhythmias);
* evidence of varices (venous insufficiency stage ≥ C2, "varicose veins");
* known abdominal aortic aneurism;
* indwelling catheterisation;
* recent surgery (3 months) requiring anaesthesia;
* known or suspected pregnancy;
* breast-feeding female participants.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on mean BP change (mmHg) after 3rd minute of head-up tilt test with respect to baseline. | 3 days

SECONDARY OUTCOMES:
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on systolic BP change (mmHg) after 3rd minute of head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on diastolic BP change (mmHg) after 3rd minute of head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on mean BP change (mmHg) after 10th minute of head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on systolic BP change (mmHg) after 10th minute of head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on diastolic BP change (mmHg) after 10th minute of head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on absolute mean orthostatic BP value (mmHg) after 3rd minute of head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on absolute systolic orthostatic BP value (mmHg) after 3rd minute of head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on absolute diastolic orthostatic BP value (mmHg) after 3rd minute of head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on absolute mean orthostatic BP value (mmHg) after 10th minute of head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on absolute systolic orthostatic BP value (mmHg) after 10th minute of head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on absolute diastolic orthostatic BP value (mmHg) after 10th minute of head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on OH symptom severity after 3rd minute of head-up tilt test with respect to baseline. | 3 days
  OH symptom severity measured by the "Orthostatic Hypotension Questionnaire (OHQ)" subcale "Orthostatic Hypotension Symptom Assessment" item-#1 [Range: 0 (minimum, i.e. "no symptoms") to 10 (maximum, i.e. "worst possible symptoms")]
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on OH symptom severity after 10th minute of head-up tilt test with respect to baseline. | 3 days
  OH symptom severity measured by the "Orthostatic Hypotension Questionnaire (OHQ)" subcale "Orthostatic Hypotension Symptom Assessment" item-#1 [Range: 0 (minimum, i.e. "no symptoms") to 10 (maximum, i.e. "worst possible symptoms")]
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on mean BP change (mmHg) after 3rd minute of active standing test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on systolic BP change (mmHg) after 3rd minute of active standing test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on diastolic BP change (mmHg) after 3rd minute of active standing test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on absolute mean orthostatic BP value (mmHg) after 3rd minute of active standing test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on absolute systolic orthostatic BP value (mmHg) after 3rd minute of active standing test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on absolute diastolic orthostatic BP value (mmHg) after 3rd minute of active standing test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on OH symptom severity after 3rd minute of active standing test with respect to baseline. | 3 days
  OH symptom severity measured by the "Orthostatic Hypotension Questionnaire (OHQ)" subcale "Orthostatic Hypotension Symptom Assessment" item-#1 [Range: 0 (minimum, i.e. "no symptoms") to 10 (maximum, i.e. "worst possible symptoms")]
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on supine mean BP value (mmHg) at 10th minute before head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on supine systolic BP value (mmHg) at 10th minute before head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on supine diastolic BP value (mmHg) at 10th minute before head-up tilt test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on supine mean BP value (mmHg) at 5th minute before active standing test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on supine systolic BP value (mmHg) at 5th minute before active standing test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on supine diastolic BP value (mmHg) at 5th minute before active standing test with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on in-lab sensor-based mean gait velocity with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus a placebo binder for two hours on in-lab sensor-based mean stride length with respect to baseline. | 3 days
Effect of wearing an elastic abdominal binder versus no binder for five consecutive days on lowest systolic BP values (mmHg) after 3rd minute of home active standing test in the early morning. | 10 days
Effect of wearing an elastic abdominal binder versus no binder for five consecutive days on lowest systolic BP values (mmHg) after 3rd minute of home active standing test 60 minutes after lunch. | 10 days
Effect of wearing an elastic abdominal binder versus no binder for five consecutive days on highest supine systolic BP values (mmHg) at 5th minute before home active standing test in the evening. | 10 days
Effect of wearing an elastic abdominal binder versus no binder for five consecutive days on OH symptom severity. | 10 days
  OH symptom severity measured by the "Orthostatic Hypotension Questionnaire (OHQ)" [Range: 0 (minimum, i.e. "no symptoms") to 100 (maximum, i.e. "worst possible symptoms")], including subcales "Orthostatic Hypotension Symptom Assessment" [Range: 0 (minimum, i.e. "no symptoms") to 60 (maximum, i.e. "worst possible symptoms")] and "Orthostatic Hypotension Daily Activitiy Scale" [Range: 0 (minimum, i.e. "no interference") to 40 (maximum, i.e. "total interference")], as well as single-item scores [Range: 0 (minimum, i.e. "no symptoms/interference") to 10 (maximum, i.e. "worst possible symptoms/total interference")]
Effect of wearing an elastic abdominal binder versus no binder for five consecutive days on overall mobility. | 10 days
  Overall mobility measured by the International Physical Activity Questionnaire (IPAQ), indicated in total physical activity metabolic equivalent minutes per week (i.e. total MET-minutes/week) [Range: 0 (minimum, i.e. "no physical activity"), no maximum (i.e. the higher the better the overall mobility)]
Effect of wearing an elastic abdominal binder versus no binder for five consecutive days on PAM-derived number of walking bouts. | 10 days
Effect of wearing an elastic abdominal binder versus no binder for five consecutive days on PAM-derived duration of walking bouts. | 10 days
Effect of wearing an elastic abdominal binder versus no binder for five consecutive days on PAM-derived mean gait velocity. | 10 days
Effect of wearing an elastic abdominal binder versus no binder for five consecutive days on PAM-derived mean stride length. | 10 days
Number of participants with treatment-related adverse events. | 8 days
  Adverse event rates will be coded by body system and MedDRA classification terms. Adverse events will be tabulated by treatment group and will include the number of participants for whom the event occurred, the rate of occurrence, the severity and relationship to the investigational medical device.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

REFERENCES:
- [Background] Fanciulli A, Goebel G, Metzler B, Sprenger F, Poewe W, Wenning GK, Seppi K. Elastic Abdominal Binders Attenuate Orthostatic Hypotension in Parkinson's Disease. Mov Disord Clin Pract. 2015 Nov 27;3(2):156-160. doi: 10.1002/mdc3.12270. eCollection 2016 Mar-Apr. PMID 30363559
- [Background] Fanciulli A, Wenning GK. Multiple-system atrophy. N Engl J Med. 2015 Jan 15;372(3):249-63. doi: 10.1056/NEJMra1311488. No abstract available. PMID 25587949
- [Background] Fanciulli A, Leys F, Falup-Pecurariu C, Thijs R, Wenning GK. Management of Orthostatic Hypotension in Parkinson's Disease. J Parkinsons Dis. 2020;10(s1):S57-S64. doi: 10.3233/JPD-202036. PMID 32716319